CLINICAL TRIAL: NCT00170274
Title: Prevention and Automatic Therapy of Atrial Arrhythmias in Patients With Paroxysmal Supraventricular Tachycardias Who Need Cardiac Pacing
Brief Title: APART: Prevention and Automatic Therapy of Atrial Arrhythmias in Patients With Paroxysmal Supraventricular Tachycardias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEN_G_CA_5
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2018-01

CONDITIONS: Tachyarrhythmia
Keywords: Indication for cardiac pacing; Atrial Arrhythmia; Indication for the implantation of a pacemaker according to the German guidelines; Documented (ECG) atrial tachyarrhythmia within the last three months before enrollment
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (No Intervention): Algorithms for prevention and termination of AF not activated
- Prevention and Therapy Algorithms on (Active Comparator): Activation of preventive and therapeutic algorithms
  Interventions: Device: Activation of preventive and therapeutic algorithms for treatment of AF; Device: AF Prevention and Therapy Algorithms On

INTERVENTIONS:
Device: Activation of preventive and therapeutic algorithms for treatment of AF — Algorithms in At 500 or Enrhyhtm for prevention and termination of Atrial Fibrillation
  Arms: Prevention and Therapy Algorithms on
Device: AF Prevention and Therapy Algorithms On — Activation of AF-prevention and termination algorithms in AT 500 or EnRhyhtm
  Arms: Prevention and Therapy Algorithms on

SUMMARY:
The goal of APART is the assessment of the therapeutic and preventive stimulation algorithms of the Medtronic AT500 and following devices in patients with atrial tachyarrhythmias and an indication for cardiac pacing according to the German guidelines. Medication is controlled throughout the study with a beta-blocker as the only antiarrhythmic drug.

ELIGIBILITY:
Inclusion Criteria:

* Indication for cardiac pacing according to the German guidelines
* Documented (electrocardiogram; ECG) atrial arrhythmia during the last three months before enrollment
* Willingness to terminate antiarrhythmic drugs until the first recurrence of an atrial arrhythmia
* Sinus rhythm during 24 hours before implant of the device

Exclusion Criteria:

* Ejection fraction below 40%
* Mechanic prosthesis of the tricuspid valve
* Indication to implantable cardioverter defibrillator (ICD)-implantation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2000-08; Primary Completion 2011-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic and/or persistent re-occurrences of atrial arrhythmias | 2 years
Time to first re-occurrence of first symptomatic or persistent atrial arrhythmia | 2 years

SECONDARY OUTCOMES:
Atrial fibrillation (AF)-burden | 2 years
Time interval between persistent episodes during the follow-up period | 2 years
Reduction of the total amount of tachyarrhythmias stored in the event counter of the implanted device | 2 years
Quality of life | 2 years
Necessity and date of a specific antiarrhythmic therapy and/or prescription of antiarrhythmic drugs class I and II | 2 years
Evaluation of possible atrial proarrhythmic effects of the termination algorithms | 2 years
Cost-efficiency | 2 years
Incidence in different pacing modes [AAI, DDD(R)] | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Wiegand, MD, Principal Investigator — Universitätsklinik Lübeck Schleswig-Holstein, Campus Lübeck; Christian Wolpert, MD, Principal Investigator — Universitätsklinik Mannheim
Locations (6):
- Germany (6):
  - Segeberger Kliniken, Bad Segeberg
  - Kath. Krankenhausgemeinschaft GmbH, Philippusstift Essen, Essen
  - Krankenhaus Marienhof, Koblenz
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Universitätsklinik Lübeck Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinik Mannheim, Mannheim

IPD SHARING:
Plan to Share IPD: No